CLINICAL TRIAL: NCT07128355
Title: A Pilot Study of Botensilimab and Balstilimab and SBRT in Non-MSI-H or pMMR Colorectal Cancer With Liver Metastasis
Brief Title: Botensilimab, Balstilimab, and SBRT in Colorectal Cancer
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Principal Investigator, Aparna Parikh, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-495
Record Dates: First submitted 2025-08-13; First posted 2025-08-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Non-MSI-H or pMMR Colorectal Cancer With Liver Metastasis
Keywords: colorectal cancer; colorectal cancer with liver metastasis; Non-MSI-H or pMMR Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiosurgery; balstilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Stereotactic Body Radiation Therapy (SBRT) + Botensilimab + Balstilimab (Experimental): Participants will receive:
  * standard of care (SOC) SBRT for 2-3 weeks (Cycle 1)
  * botensilimab, on Day 1 of 6-week cycles (Cycles 1-4)
  * balstilimab, once every 2 weeks (Cycles 1-14, 6-week cycles)
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Drug: Botensilimab; Drug: Balstilimab

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Starting on Day 1 participants will have 2-4 treatments per week for about 2 weeks, with no more than 2 days in a row. This is expected to last about 2 weeks but could last up to 3 weeks.
  Other Names: SBRT
Drug: Botensilimab — Administered once every 6 weeks by intravenous infusion over about 30 minutes, on Day 1 of Cycles 1-4 (six-week cycles). Administered 30 minutes after balstilimab.
  Other Names: AGEN1181
Drug: Balstilimab — Administered once every 2 weeks by intravenous infusion over about 30 minutes, starting on Day 1 of Cycle 1 and continuing for 4 six-week cycles (with botensilimab) followed by up to 14 six-week cycles of balstilimab alone. Participants will receive balstilimab for a total of 18 six-week cycles.
  Other Names: AGEN2034

SUMMARY:
This is a single-arm pilot feasibility study evaluating the combination of Botensilimab and Balstilimab with Radiation Therapy (RT) in Non-Microsatellite Instability High (MSI-H) or Proficient Mismatch Repair (pMMR) chemorefractory colorectal cancer (CRC) with liver metastasis.

DETAILED DESCRIPTION:
In this open-label study, the investigators propose to use standard of care (SOC) radiation (Stereotactic Body Radiation Therapy (SBRT)) to control the liver lesions in combination with investigational dual checkpoint inhibitors, botensilimab (AGEN1181) and balstilimab (AGEN2034).

Initially, 5 patients will be enrolled in a lead-in cohort and assessed for dose-limiting toxicity (DLT) related to radiation during Cycle 1. If DLT are observed in 2 or more of the first 5 patients, the protocol will be stopped early. If DLT were observed in 0 or 1 of the first 5 patients during the lead-in, enrollment will be expanded to a total of 15 patients. After screening, participants will receive SOC SBRT for 2-3 weeks, and botensilimab + balstilimab for up to 24 weeks followed by balstilimab alone for 14 additional 6-week cycles, for a total treatment time of up to 108 weeks. Participants will be followed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed adenocarcinoma of colorectal origin.
* MSI-H or pMMR status confirmed by IHC or PCR.
* Must have at least 1 measurable (≥ 1 cm) previously unirradiated hepatic lesion amenable to ablative RT and can meet dose constraints; maximum 5 lesions are allowed given each lesion is no larger than 3 cm. Must have at least 1 other unirradiated measurable (≥ 1cm) extrahepatic lesion, outside of RT field. Must have at least 700 cc of unaffected liver.
* Must have received or confirmed intolerance to 5-FU, Oxaliplatin, and Irinotecan (in any combination).
* Age ≥18 years
* ECOG performance status ≤ 1
* Life expectancy of greater than 3 months.
* Participants must meet the following organ and marrow function as defined below:

  * Absolute Neutrophil Count (ANC) ≥ 1500 /mcL
  * White Blood Cells (WBC) ≥ 2000 /mcL
  * Platelets (PLT) ≥ 100,000 /mcL
  * Hemoglobin (HGB) ≥ 8 g/dL without transfusion within 2 weeks of measurement
  * AST and ALT ≤ 2.5 x ULN
  * Total Bilirubin ≤ 1.5 x ULN OR < 3 mg/dL for participants with Gilbert Syndrome
  * Creatinine Clearance ≥ 40 mL/min if calculated using Cockcroft-Gault formula
* The effects of radiation on the developing human fetus are known to be teratogenic and the safety of Botensilimab and Balstilimab in pregnant women and their fetuses has not been established.

  --Woman of childbearing potential (WOCBP) and men with WOCBP partners must agree to use highly effective contraceptive measures starting at screening through 5 months (180 days) after the last dose of balstilimab and/or botensilimab.
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG).
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy, targeted small molecule therapy or study therapy within 14 days prior to starting protocol treatment, or those who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 2 weeks earlier.

  * EXCEPTION: Participants with ≤ Grade 2 neuropathy are permitted.
  * If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting protocol treatment.
* Known or suspected, active, autoimmune disease
* Condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to study drug administration.

  --EXCEPTIONS: Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if >10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* Positive TB (Bacillus Tuberculosis) at screening. NOTE: skin test is not allowed. Interferon-Gamma Release Assay (IGRA)-based tests such as QuantiFERON TB Gold and T-Spot TB tests are acceptable.
* Partial or complete bowel obstruction within the last 3 months, signs/ symptoms of bowel obstruction, or known radiologic evidence of impeding obstruction.
* Refractory ascites defined as requiring 2 or more therapeutic paracenteses within the last 4 weeks, or ≥ times within the last 90 days, or ≥ time within the last 2 weeks prior to study entry, or requiring diuretics within 2 weeks of study entry.
* Known history of active or chronic HBV or HCV infection
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). These participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.

  -- EXCEPTIONS: Patients with CD4 >200 cells/mm3 and/or undetectable viral load are eligible.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Participant is pregnant, breastfeeding, expecting to conceive, or father children within the projected duration of the trial, starting with the consent visit through 120 days for woman and 120 days for men, after the last dose of study treatment.

There is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with radiation, breastfeeding should be discontinued if the mother is treated with radiation.

* Known history of, or any evidence of active, non-infectious pneumonitis.
* Active infection requiring systemic therapy.
* Has received a live vaccine within 30 days of planned start of study therapy. Intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

  --EXCEPTION: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to any study agents.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Uncontrolled brain metastases. Participants treated with radiation > 4 weeks prior to registration, with follow up imaging showing control are eligible.
* Participants who present with significant active diarrhea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting radiation-related toxicities | Day 1 of treatment through 30 days after completion of radiation therapy (radiation therapy is 2-3 weeks), up to 60 days.
  Dose limiting radiation-related toxicities will be assessed by CTCAE v5.0. A dose limiting toxicity (DLT) will be defined as any patient who can't complete all radiation therapy (RT) fractions within 2-3 weeks for pre-specified toxicity or lab values attributable to radiation therapy, or development of RT-related toxicities within 30 days of completion of RT. Participants will be evaluable for DLT once they start protocol therapy.

SECONDARY OUTCOMES:
Response rate of in-field radiated hepatic lesion(s) | Screening through end of Cycle 18 (each cycle is 6 weeks), up to 108 weeks.
  The response rate (Complete Response (CR), Partial Response (PR)) of irradiated hepatic lesions by RECIST 1.1 will be estimated as a proportion with 95% confidence intervals based on the exact binomial distribution by RECIST.
Response rate of extrahepatic lesion(s) | Screening through end of Cycle 18 (each cycle is 6 weeks), up to 108 weeks.
  The response rate (Complete Response (CR), Partial Response (PR)) of unirradiated extrahepatic lesions by RECIST 1.1 will be estimated with 95% confidence intervals based on the exact binomial distribution.
Overall Survival (OS) | Registration through 160 weeks (108 weeks of treatment + 1 year follow-up)
  OS is defined as time from registration to death due to any cause or censored at date last known alive. OS rates will be estimated using the Kaplan-Meier method with 95% confidence intervals based on the complementary log-log transformation.
Progression-Free Survival (PFS) | Registration through up to 108 weeks of treatment
  PFS is defined as time from registration to the earlier of progression (per RECIST 1.1) or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation. PFS rates will be estimated using the Kaplan-Meier method with 95% confidence intervals based on the complementary log-log transformation.
Disease Control Rate (DCR) | Day 1 through up to 108 weeks.
  Disease control is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements. Response is measured by RECIST 1.1. The cumulative incidence will be estimated with patients still alive with disease control censored at the date of last disease assessment and death without disease analyzed as a competing risk.

CONTACTS AND LOCATIONS:
Overall Officials: Aparna R. Parikh, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to the PI, Aparna Raj Parikh, MD, MS (aparna.parikh@mgh.harvard.edu). The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation